CLINICAL TRIAL: NCT06119620
Title: Brain Outcome After Cardiac Arrest. Modifying Working Memory With Non-invasive Brain Stimulation - A Series of SCEDs
Brief Title: Modifying Working Memory With Brain Stimulation
Acronym: BROCA-NIBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BROCA-NIBS
Record Dates: First submitted 2023-10-26; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Arrest; Cognitive Impairment
MeSH Terms: conditions — Heart Arrest; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a single case experimental design. All participants will receive both sham and active stimulation. The order of stimulation (sham, active, sham active OR active, sham, active, sham) will be randomised. Also the length of the N-back task is randomised between 8, 10, and 12 minutes).
Masking Description: The participant won't be told if they receive sham or active stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABAB (Other): all participants will go through sham (control) and active (experimental) stimulation. So either sham - active - sham - active or active - sham - active - sham
  Interventions: Device: intermitted theta burst stimulation

INTERVENTIONS:
Device: intermitted theta burst stimulation — Participants receive intermitted theta burst stimulation for 3-4 minutes before completing the N-back task.
  Other Names: rTMS

SUMMARY:
The investigators want to investigate the effect of rTMS on working memory measured by the N-back task. This is a single case experimental design, ABAB.

DETAILED DESCRIPTION:
Rationale: The survival rate of patients after cardiac arrest and resuscitation has increased considerably. A common consequence of cardiac arrest is ischemic-hypoxic brain damage leading to cognitive impairment. Currently, there is a lack of knowledge regarding effectiveness of treatments to improve outcomes of patients with cognitive impairment after a cardiac arrest.

Objective: The primary objective is to investigate the effects of rTMS (iTBS protocol) on working memory of people with memory impairments after a cardiac arrest in the past Study design: This will be a single blinded replicated randomized SCED withdrawal designs study.

Study population: Nine adults who had a cardiac arrest in the past will be participating in this study. They are recruited in the general population.

Intervention: If participants are suitable based on the screening. Participants are invited to the university of Maastricht. There they receive intermitted theta burst stimulation with a TMS coil for 3 minutes on the dorsolateral prefrontal cortex. Then they perform the N-back task for 8 to 12 minutes to estimate working-memory performance. Then they have a break (45 min). Then they receive 3 minutes of sham stimulation after which they have to perform the N-back task again for 8 - 12 minutes. This will be repeated (active stimulation - sham - active stimulation - sham).

Main study parameter: The main study outcomes are performance on the N-back task with regard to accuracy.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The participant has to come to the university twice. The screening session takes approximately 1-1,5 hour, the experimental session 3,5 hours. The participant could experience side effects of the rTMS, these include: headache, scalp discomfort, tingling or twitching of the facial muscles, and light-headedness. Serious side effects are very rare, but they may include: seizures. The N-back task can be experienced as tiring.

ELIGIBILITY:
Inclusion Criteria:

* Had a cardiac arrest between 3 months and 5 years prior to the experiment session.
* Scores lower than the general population (corrected for age, education, and sex) on at least one of the cognitive tests ( SD < -1 on the Stroop, digit span, or TMT).
* Age 18 up to and including 75.
* Proficient in Dutch or English to understand the instructions for the N-back task.
* Has sufficient understanding to perform the N-back task.
* Written informed consent

Exclusion Criteria:

* Has a pacemaker or ICD (implantable cardioverter-defibrillator)
* A history or a family member with a history of seizures / epilepsy (asked on the phone and checked on the first appointment).
* Metal implants in or near the head.
* Pregnancy
* Any other neurological disorder impending working memory performance besides the OHCA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy on the N-back task | 1 measurements every 2 minutes for 8 - 10 minutes after each N-back task (4 times in total)
  Percentage of correct responses for every 2 N-back blocks

SECONDARY OUTCOMES:
RT on the N-back task | 1 measurements every 2 minutes for 8 - 10 minutes after each N-back task (4 times in total)
  reaction time on the N-back task
d' on the N-back task | 1 measurements every 2 minutes for 8 - 10 minutes after each N-back task (4 times in total)
  d' = z(False alarms) - z(Hits)

CONTACTS AND LOCATIONS:
Overall Officials: Caronline v van Heugten, Dr. prof., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No